CLINICAL TRIAL: NCT06119997
Title: Screening for Advanced Liver Fibrosis Using Non-invasive Tests in Primary Care
Acronym: ANTICIP-SP
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC22.0266
Record Dates: First submitted 2023-10-12; First posted 2023-11-07 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Hepatic Fibrosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Liver fibrosis screening is possible at the asymptomatic stage through a healthcare management strategy currently recommended for patients with risk factors for chronic liver disease. It is based on a sequential strategy involving a 1st-line test, fibrosis score calculation (FIB-4).

Given this opportunity to identify advanced fibrosis in asymptomatic patients, the project aims to set up this screening program in the Grenoble area with Biogroup Laboratories, in collaboration with the Hepato-gastroenterology department (HGE) of Grenoble University Hospital. The aim of this study is to evaluate the success of sequential screening using FIB-4, followed by a specialized fibrosis test for the diagnosis of advanced hepatic fibrosis

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 70 years of age
* FIB-4 2.67
* Patients covered by Health Insurance System

Exclusion Criteria:

* Prescription triggering FIB-4 emanate from a hepatogastroenterologist or oncologist
* Conditions associated with high risk false-positive FIB-4: ASAT or ALAT > 300 IU/L, platelets <50 G/L or >500 G/L.
* Patient refusing to participate
* Subjects under guardianship or deprived of liberty

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study Population (FIB-4 ≥2.67):
  The expected frequency of advanced fibrosis in the study population (= positive predictive value) is estimated at 14%, based on literature data (sensitivity and specificity of FIB-4 ≥2.67 for the diagnosis of advanced fibrosis at 32% and 96%, prevalence of advanced fibrosis at 2% in the screened population (10)). Assuming adherence to recommendations to achieve a 10% diagnosed liver fibrosis, corresponding to a non-inferiority margin of 4% compared to the theoretical percentage of 14%, 441 patients are required (power at 80%, alpha risk at 5%, binomial test for a single sample). This sample size will be extended to 500 patients with FIB-4 ≥2.67, taking potential attrition into account.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the sequential screening of advanced hepatic fibrosis in primary care using an automatic calculation of FIB-4 followed by the use of a specialized non-invasive fibrosis test | up to 14 months
  Percentage of patients with advanced hepatic fibrosis (fibrosis at least equivalent to stage F3 or F4 according to METAVIR at the end of the evaluation by the hepatogastroenterologist) diagnosed among patients with no known HCV infection and FIB-4 ≥2.67
Evaluation of diagnoses of advanced hepatic fibrosis made during the study compared to the expected disease frequency | up to 14 months
  Proportion of diagnoses made at 14 months to the expected disease frequency among patients with no known HCV infection and FIB-4 ≥2.67

SECONDARY OUTCOMES:
Among all patients with calculated FIB-4 scores, evaluate the proportion of patients eligible for a specialized hepatic fibrosis assessment test. | up to 12 months
  Proportion of patients with FIB-4 ≥2.67 among patients who underwent FIB-4 calculation or the screened population.
Evaluate, among patients with FIB-4 ≥2.67, the proportion of pathways compliant at 14 months. | up to 14 months
  Proportion among patients with FIB-4 ≥2.67 who have received appropriate medical care, defined by the performance of a specialized test and a specialist consultation if the test is positive.
Evaluate, among patients diagnosed with advanced fibrosis, the proportion of specialized follow-ups compliant with recommendations at 14 months. | up to 14 months
  Proportion among patients with advanced fibrosis who have had at least one specialist consultation, and for patients with cirrhosis, a semi-annual screening ultrasound for HCC within 14 months.
Description of social and clinical determinants associated with the diagnosis of advanced fibrosis and the quality of follow-up at 14 months | up to 14 months
  Estimation of crude and adjusted relative risks for advanced liver fibrosis and non-compliant follow-up associated with the following variables: age, sex, smoking, diabetes, obesity, sleep apnea syndrome, high blood pressure, dyslipidemia, alcohol consumption, screening for alcohol-related risks, physical activity, medical history, current treatments, level of education, socio-professional category, assessment of precariousness, existence of situations of non-use of healthcare